CLINICAL TRIAL: NCT04605887
Title: Angiotensin 1-7 as a Therapy for Pneumonia Caused by Coronavirus 2(SARS-CoV-2)
Brief Title: Angiotensin 1-7 as a Therapy in the Treatment of COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Constant Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0328-20-RMB; MOH_2020-11-02_009463 (Other: Ministry Of Health Israel)
Record Dates: First submitted 2020-10-27; First posted 2020-10-28 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — angiotensin I (1-7)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Active Comparator): Ang 1-7 subcutaneously 500 mcg/kg /day
  Interventions: Drug: Angiotensin 1-7
- control group (Placebo Comparator): NaCl 0.9% subcutaneously 2.0 cc once a day
  Interventions: Drug: Angiotensin 1-7

INTERVENTIONS:
Drug: Angiotensin 1-7 — Ang 1-7 subcutaneously 500 mcg/kg /day

SUMMARY:
Phase 2 ,double blind, randomized study of therapy with Angiotensin 1-7 in COVID-19 patients. 120 confirmed SARS-CoV-2 infected patients who exhibit moderate- clinical symptoms including dyspnea, cough and fever, hospitalized in the KETER department in several hospitals in Israel, will be enrolled. 60 patients will receive Ang 1-7 subcutaneously 500 mcg/kg /day. 60 patients will receive placebo : NaCl 0.9% 2 ml -control arm .

Treatment duration: 14 days or until clinical improvement that enables discharge from hospital.

(the shortest time will be the limiting factor in treatment duration). Follow-up-30 days. 14-30 days after discharge from hospital: we will contact the patient via phone to ask questions related to any possible adverse reaction to the drug and general health.

DETAILED DESCRIPTION:
The working hypothesis behind this study is that the deleterious effects of SARS-CoV-2 are largely attributed to the deprivation of the affected target cells from their advantageous ACE-2-Ang 1-7-MasR machinery on one hand, and to the use of ACE2 as a Trojan horse to infect and destroy these cells on the other in a vicious feed-forward cycle.

120 confirmed SARS-CoV-2 infected patients who exhibit moderate- clinical symptoms including dyspnea, cough and fever, hospitalized in the KETER department in several hospitals in Israel, will be enrolled. 60 patients will receive Ang 1-7 subcutaneously 500 mcg/kg /day. 60 patients will receive placebo : NaCl 0.9% 2 ml -control arm .

Treatment duration: 14 days or until clinical improvement that enables discharge from hospital.

All patients will be treated by Dexamethasone and Remdesivir, according to the published guidelines. Moreover, if other promising medications will be approved for COVID-19, the patients will also be treated by these medications. The current trial will not exclude promising COVID-19 treatments.

Each patient will be closely followed up, where routine physical sings, respiratory and hemodynamic parameters will be documented. In addition, the following complications will be monitored: thromboembolic events, myocarditis, impaired liver function and acute kidney injury. Allergic reactions will be treated by corticosteroids, antihistamines and adrenalin if needed. Patients experiencing allergic reactions will be excluded from continuing the trail.

In addition, biochemical (kidney function tests, electrolytes, liver enzymes, albumin, protein, ferritin, troponin- 5 ml) and hematological (CBC-(3 ml), and coagulation tests-(3 ml)) analysis will be performed on the day of enrollment and every 3 days . Other blood tests for immunophenotyping, cytokines, COVID-19 PCR, Angiotensin II (Ang II) levels, Angiotensin 1-7 (Ang 1-7) levels, ACE and ACE-2 will be collected at baseline and at days 6,15,21 and 30 days after enrollment. and every week ( 2 chemistry (10 ml) and 2 CBC tubes (10 ml)).

In addition chest X-ray will be performed at enrollment and at days 6,15,21 and 30 days after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Respiratory specimen is positive for SARS-CoV-2 nucleic acid by RT-PCR
2. Fever: Temperature >37.8℃
3. Moderate lung disease, defined by the following respiratory variables (meets one of the following criteria): lung infiltrates (evident by chest X-ray) not attributable to other causes plus one of the following:

   * Respiratory rate: RR ≥25 breaths/min
   * Oxygen saturation ≤94 % at rest on room air
4. HBsAg negative, HCV negative; HIV negative
5. Informed consent

   -

   Exclusion Criteria:
   * Age <18 years
   * Pregnant or breast-feeding woman or with positive pregnancy test result
   * PaO2/FiO2 ≤100 mmHg / mechanical ventilation
   * Severe organ failure - not expected to survive for >7 days
   * Hemodynamically unstable in the preceding 10 hours (MAP ≤65 mmHg, or SAP <90 mmHg, DAP <60 mmHg, vasoactive agents are required)
   * Patient on ECMO
   * Patient in other therapeutic clinical trial within 30 days before enrolment
   * Chronic immunosuppression: current autoimmune diseases or patients who received immunotherapy within 30 days before enrolment
   * Hematologic malignancy (lymphoma, leukemia, multiple myeloma)
   * Other patient characteristics (not thought to be related to underlying COVID-19) that portend a very poor prognosis (e.g, severe congestive heart failure( NYHA class III or IV, EF less than 30%,) liver cirrhosis , chronic kidney disease stave IV, V(e GFR<30 ml/min), chronic obstructive lung disease: GOLD C,D : ≥2 exacerbations or ≥1 that required hospitalization, FEV1<50%, GOLD 3,4)
   * Atopic patients suffering from allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Need for mechanical ventilation | Any time from randomization up to 30 days of last study treatment dose
  Patient is intubated
Death | Any time from randomization up to 30 days of last study treatment dose
  death certificate

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No